CLINICAL TRIAL: NCT00896155
Title: A Randomized Trial of Concurrent Versus Sequential Tamoxifen With Radiotherapy to Assess the Extent of Pulmonary Fibrosis and Disease Related Control and Survival in Breast Cancer Patients
Brief Title: Trial of Concurrent Versus Sequential Tamoxifen With Radiotherapy in Breast Cancer Patients
Acronym: CONSET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Anusheel Munshi, Associate Professor, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 349
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Pulmonary Fibrosis; Breast Cancer
Keywords: Breast cancer; Pulmonary fibrosis; tamoxifen; radiotherapy
MeSH Terms: conditions — Pulmonary Fibrosis; Breast Neoplasms | interventions — Tamoxifen; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concurrent Tamoxifen and Radiotherapy (Experimental): ARM 1 will receive Tamoxifen given concurrently with radiotherapy. Tamoxifen will continue for a period of 5 years.
  Interventions: Drug: Tamoxifen; Radiation: Radiotherapy
- Sequential radiotherapy and tamoxifen (Active Comparator): ARM-2 shall receive radiotherapy followed by tamoxifen sequentially. Again tamoxifen will continue for a period of 5 years.
  Interventions: Drug: Tamoxifen; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Tamoxifen — 260 patients of breast cancer will be accrued into the study. After inclusion in the study, all the patients will be randomized into two arms. ARM 1 will receive Tamoxifen 20 Mg once daily given concurrently with radiotherapy while in ARM-2 radiotherapy followed by tamoxifen 20 mg once daily sequentially.
Radiation: Radiotherapy — 260 patients of breast cancer will be accrued into the study. After inclusion in the study, all the patients will be randomized into two arms. ARM 1 will receive Tamoxifen 20 Mg once daily given concurrently with radiotherapy while in ARM-2 radiotherapy followed by tamoxifen 20 mg once daily sequentially.

SUMMARY:
Two hundred and sixty patients with breast cancer will be accrued into the study. After inclusion in the study, all the patients will be randomized into two arms. Arm 1 will receive Tamoxifen given concurrently with radiotherapy while in Arm 2 radiotherapy will be given followed by tamoxifen sequentially. The patients will be stratified for the following factors: a) BCS (Breast conservative surgery) versus MRM (modified radical mastectomy) and b) central lung distance (CLD) > 2 cm.

Patients in both arms will continue tamoxifen for a period of 5 years. The patients will be evaluated by high-resolution computed tomography (HRCT) (baseline and at 2 years), serum transforming growth factor (TGF) beta levels (baseline and at 6 months) and diethylenetriaminepentaacetic acid (DTPA) aerosol clearance half life (baseline and at 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients with large operable lesions (pT/cT > 5 cm) or locally advanced breast cancers undergoing modified radical mastectomy or breast conservative surgery-(BCS) who need adjuvant post operative radiotherapy
* Patients post mastectomy requiring radiotherapy because of nodal positivity
* Completed planned chemotherapy schedule
* ER and/or PR positive patients
* Patients decided to be put on tamoxifen
* Patients reliable for follow up

Exclusion Criteria:

* Patients with BCT who have pT1 or pT2 breast lesions (N0,N1)
* Patients for palliative radiotherapy to the chest wall/breast/supraclavicular fossa
* Any patient requiring radiation to the axillary or internal mammary area
* Recurrent disease or metastatic disease
* Patients on concurrent chemotherapy and radiation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Development of Lung fibrosis | Three years

SECONDARY OUTCOMES:
Locoregional failure and distant failure | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Anusheel Munshi, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Center, Pārel, Mumbai, India